CLINICAL TRIAL: NCT07347873
Title: Diagnostic Accuracy of the Clinical Tests and the Musculoskeletal Ultrasonography in Lateral Elbow Tendinopathy
Brief Title: Diagnostic Accuracy of the Clinical Tests and the Ultrasonography in Lateral Elbow Tendinopathy
Status: Recruiting | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, İlker Yağcı, Prof. M.D., Marmara University
Other Study IDs: 09.2025.25-0880
Record Dates: First submitted 2025-12-24; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Lateral Elbow Tendinopathy (Tennis Elbow)
Keywords: Elbow pain; Lateral epicondylitis; Cozen; Elastography
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lateral elbow tendinopathy: Patients with lateral epicondylitis will be included in this group.
- Control: Healthy volunteers with similar demographic characteristics will be enrolled to this group.

SUMMARY:
Lateral elbow tendinopathy (LET) is the most common cause of elbow pain. Even though provocation tests such as Cozen's test, Mill's test or Maudsley test; musculoskeletal ultrasound or magnetic resonance imaging can be used for diagnosis, gold standard method is yet to be determined. Purpose of this study is to determine the sensitivity and specificity of clinical tests and ultrasonography in diagnosis of LET.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-60 with unilateral elbow pain
* Tenderness with palpation at the lateral epicondyle
* Pain triggered with pressure compared to the opposite lateral epicondyle with algometer.

Exclusion Criteria:

* History of rheumatologic diseases
* History of e corticosteroid injections on lateral epicondyle
* History of elbow surgery or infection

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients presented to the outpatient clinic of Physical Medicine and Rehabilitation of Marmara University with elbow pain and diagnosed with lateral epicondylitis will be informed about the study. Willing patients will be enrolled after written consent is taken.
  Control group will be chosen with volunteers, which have similar demographic characteristics.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-10-17 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-03-26 (Estimated)

PRIMARY OUTCOMES:
Elastography | At enrollment
  Both shear wave and strain elastography will be applied. Stiffness and shear wave velocity will be calculated on shear wave elastography and strain ratio will be calculated on strain elastography.

SECONDARY OUTCOMES:
Musculoskeletal ultrasound | At enrollment
  Sonographic evaluation will begin with gray scale examination. Swelling, cortical irregularity, hypoechogenicity, calcification, tear common extensor tendon thickness will be assessed. Power doppler will be evaluated between the superficial fibers of the common extensor tendon, the bone surface, the insertion point of the common extensor tendon and the humeroradial joint. Doppler activity will be graded based in a 0.5-cm longitudinal part of the tendon with the maximal Doppler activity (the region of interest-ROI). The 5-point grading will be as follows. Grade 0: No activity, Grade 1: Single vessel, Grade 2: Doppler activity in 0-25% of the ROI, Grade 3: Doppler activity in 25-50% of the ROI, Grade 4: Doppler activity in >50 of ROI. Lastly elastography will be used.
Cozen's test | At enrollment
  Resisted wrist extension will be performed while patient is sitting and elbow on extension. Cozen's test will be applied to both extremities. Pain felt on the lateral epicondyle during provocation indicates a positive test result.
Maudsley's Test | At enrollment
  Resisted third finger extension will be performed while patient is sitting and elbow on 90 degrees flexion. Maudsley's test will be applied to both extremities. Pain felt on the lateral epicondyle during provocation indicates a positive test result.
Mill's test | At enrollment
  Maximal wrist flexion will be performed while patient is sitting, elbow on extension and forearm pronation. Mill's test will be applied to both extremities. Pain felt on the lateral epicondyle during provocation indicates a positive test result.
Hand Grip Strength | At enrollment
  Both painless and maximum grip strength will be examined using Jamar's hand dynamometer.
Algometer | At enrollment
  Force will be applied to lateral epicondyle using an algometer.
Patient Rated Tennis Elbow Evaluation | At enrollment
  Patient Rated Tennis Elbow Evaluation will be used to assess pain and functional status in patients diagnosed with LET.

CONTACTS AND LOCATIONS:
Overall Officials: İlker Yağcı, Prof. M.D., Principal Investigator — Acıbadem Ataşehir Hospital
Locations (1):
- Marmara University, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Due to legal restrictions, all data will be anonymized. Individual participant data won't be shared to third parties.

REFERENCES:
- [Background] Krogh TP, Fredberg U, Ammitzboll C, Ellingsen T. Clinical Value of Ultrasonographic Assessment in Lateral Epicondylitis Versus Asymptomatic Healthy Controls. Am J Sports Med. 2020 Jul;48(8):1873-1883. doi: 10.1177/0363546520921949. Epub 2020 Jun 2. PMID 32484714
- [Background] Hong S, Hahn S, Yi J, Park EJ, Bang JY. Comparing the clinical application of strain elastography and shear wave elastography for the evaluation of lateral epicondylitis. J Clin Ultrasound. 2023 Jan;51(1):123-130. doi: 10.1002/jcu.23356. Epub 2022 Sep 28. PMID 36169174
- [Background] Karanasios S, Korakakis V, Moutzouri M, Drakonaki E, Koci K, Pantazopoulou V, Tsepis E, Gioftsos G. Diagnostic accuracy of examination tests for lateral elbow tendinopathy (LET) - A systematic review. J Hand Ther. 2022 Oct-Dec;35(4):541-551. doi: 10.1016/j.jht.2021.02.002. Epub 2021 Feb 27. PMID 33814224